CLINICAL TRIAL: NCT00809887
Title: Micafungin Lock Therapy to Clear Fungemia While Attempting to Preserve Central Venous Catheters
Brief Title: Micafungin Lock Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to enroll subjects
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Patti Shugarts, KAI Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10882
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-11

CONDITIONS: Catheter-Related Fungal Infections
Keywords: catheter fungal infections, antimicrobial lock therapy, micafungin, central venous catheter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): ALT with placebo with systemic Micafungin therapy
  Interventions: Drug: Micafungin lock therapy
- 2 (Experimental): ALT with Micafungin and heparin with systemic Micafungin therapy
  Interventions: Drug: Micafungin lock therapy

INTERVENTIONS:
Drug: Micafungin lock therapy

SUMMARY:
The study proposes to investigate, in children admitted at Children's Medical Center at Dallas, the effectiveness of antimicrobial lock therapy (ALT) with Micafungin in combination with systemic antifungal therapy in catheter-related fungal infections in order to salvage highly needed central venous catheter (CVC) and at the same time to investigate the effectiveness of Micafungin alone as systemic therapy in the treatment of Candidemia in a pediatric population.

DETAILED DESCRIPTION:
The antimicrobial lock therapy (ALT) consists of filling a catheter lumen with a supraphysiologic concentration (100- to 1000- fold higher) of an antimicrobial agent and allowing it to dwell (lock) for several hours in an attempt to sterilize the lumen. Advantages of the ALT are: the ability to administer high local concentrations; the ease of administration; the cost-savings and vein access-savings by decreasing the number of surgical procedures in an operating room for catheter replacement; the decrease in possible surgical complications and risks. The Infectious Diseases Society of America, the Society for Healthcare Epidemiology of America and others recommend the ALT for the treatment of uncomplicated bacteremias. This technique however is not currently recommended for the treatment of catheter-related fungal infections, primarily due to lack of adequate data. This study plans to enroll approximately 20 children admitted to the Children's Medical Center at Dallas in high need of central venous catheters or with evidence of fungemia in this study to investigate the effectiveness of ALT with Micafungin against fungal infections.

ELIGIBILITY:
Inclusion Criteria:

* Children, 6 months-18 yrs, with a central line fungal infection, presumed Candida, admitted at Children's Medical Center.
* Signed informed consent by parents and assent by minor if applicable.
* Subjects with likely survival beyond 1 week.

Exclusion Criteria:

* Pocket, tunnel or exit-site infection
* Known allergic reactions to the Micafungin or echinocandins.
* Severe systemic symptoms (disseminated candidemia, fungal balls, endocarditis)
* Mixed infections
* Inability to lock the catheter lumen for minimum 8h because of other medications administration
* Subjects requiring ECMO or CVVH.
* Patients with HIV, congenital immunodeficiencies.
* Positive pregnancy test or breastfeeding.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-06 (Estimated); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Central vascular catheter preserved during lock therapy as a result of resolution of symptoms and negative cultures within 96h. | 96 hours

SECONDARY OUTCOMES:
Descriptive analysis of safety profile of patients receiving ALT and systemic micafungin | Up to one month

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center of Dallas/University of Texas Southwestern Medical Center, Dallas, Texas, United States